CLINICAL TRIAL: NCT03458416
Title: A Multicenter, Open-Label Study to Assess the Long-Term Safety of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Patients With Prader-Willi Syndrome
Brief Title: A Study to Assess the Long-Term Safety of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Participants With Prader-Willi Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insys Therapeutics filed Chapter 11 and terminated all studies.
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Collaborators: Benuvia Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS011-17-115
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabidiol Oral Solution: 20-40 mg/kg/day (Experimental): Participants will receive total daily doses between 20 milligrams per kilograms per day (mg/kg/day), 30 mg/kg/day, and 40 mg/kg/day. The two equivalent doses will be administered twice a day with a standard meal approximately every 12 hours.
  Interventions: Drug: Cannabidiol Oral Solution

INTERVENTIONS:
Drug: Cannabidiol Oral Solution — An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).

SUMMARY:
The objective of this study is to assess the long-term safety and tolerability of Cannabidiol Oral Solution (CBD) in participants with Prader-Willi Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Completed activities up to and including Visit 10 (Study Completion) of INS011-16- 085.
2. Participant and/or parent(s)/caregiver(s) fully comprehend the informed consent form and assent form, understand all study procedures, and can communicate satisfactorily with the investigator and study coordinator, in accordance with applicable laws, regulations, and local requirements.
3. If female, is either not of childbearing potential or practicing medically acceptable methods of birth control.
4. Psychotropic treatment will be permitted if the participant has been on a stable dose during the INS011-16-085 and does not anticipate a dose change during the course of the study.
5. Growth hormone treatment will be permitted if the participant has been on a stable dose during INS01-16-085.
6. Any other treatment including thyroid hormones should be stable prior to entering the INS011-17-115 study.
7. In the opinion of the investigator, the parent(s)/caregiver(s) is (are) willing and able to comply with the study procedures and visit schedules, including venipuncture, and the visit schedules.

Exclusion Criteria:

1. Participant or parent(s)/caregiver(s) have commitments during the study duration that would interfere with attending all study visits.
2. Experienced an anoxic episode related to study drug requiring resuscitation during the previous study.
3. Uncontrolled Type I and Type II Diabetes.
4. Developed an adverse event thought to be related to CBD in the previous study and the investigator determines that continuing treatment with CBD would not be in the best interest of the partient.
5. History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or other condition which would jeopardize safety or impact validity of results (per investigator).
6. Currently taking felbamate.
7. Compromised respiratory function or severe respiratory insufficiency.
8. Pregnant or lactating female.
9. In the opinion of the investigator, the participant is unsuitable in any other way to participate in this study.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkashef, MD, Study Director — INSYS Therapeutics Inc
Locations (1):
- Institute for Research and Innovation | MultiCare Health System, Tacoma, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Pre-assignment Details: Participants were enrolled in this long-term safety study after completing the INS011-16-085 study. Only 2 participants enrolled in this study. The participants received cannabidiol oral solution (CBD) doses for up to 48 weeks, and a follow-up period of 30 days.
Groups:
- Cannabidiol Oral Solution: Participants received 20 milligrams (mg)/kilogram (kg)/day to 40 mg/kg/day of CBD given twice daily with standard meals.
Period: Overall Study
Arm/Group | Cannabidiol Oral Solution
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Groups:
- Cannabidiol Oral Solution: Participants received 20 mg/kg/day to 40 mg/kg/day of CBD given twice daily with standard meals.
Arm/Group | Cannabidiol Oral Solution
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Incidence Of Adverse Events (AEs) And Serious Adverse Events (SAEs) Associated With Cannabidiol Oral Solution
Description: AE is defined as any untoward medical occurrence in a participant administered with a pharmaceutical product which does not necessarily have a causal relationship with the treatment. An SAE is defined as any event that results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or a congenital anomaly/birth defect. A summary of other non-serious AEs and all serious AEs regardless of causality, is located in the Reported AE section.
Time Frame: Up to Week 52
Population: as for baseline characteristics
Groups:
- Cannabidiol Oral Solution: Participants received total daily doses between 20 mg/kg/day to 40 mg/kg/day given twice daily with standard meals.
Arm/Group | Cannabidiol Oral Solution
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 52 Weeks
Description: This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Groups:
- Cannabidiol Oral Solution: Participants received total daily doses between 20 to 40 mg/kg/day given twice daily with standard meals.
Arm/Group | Cannabidiol Oral Solution
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT03458416/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT03458416/SAP_001.pdf